CLINICAL TRIAL: NCT06091020
Title: A Parallel-group Treatment, Proof-of-concept Phase 2, Multicenter, Double-blind, Randomized Two-arm Clinical Trial to Investigate the Efficacy and Safety of Subcutaneous NT 201 Injections Compared With Placebo Injections in Decreasing Pain Intensity in Male and Female Participants Aged 18 Years and Older With Moderate to Severe Chronic Peripheral Neuropathic Pain Due to Postherpetic Neuralgia or Peripheral Nerve Injury
Brief Title: A Clinical Trial to Investigate Efficacy and Safety of NT 201 Injections Compared With Placebo Injections in Participants Aged 18 Years and Older With Chronic Nerve Pain After Shingles or Nerve Injury
Acronym: PaiNT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Organization: Merz Pharmaceuticals GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M602011079; 2022-501461-52-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Moderate to Severe Chronic Peripheral Neuropathic Pain (PNP) Due to Postherpetic Neuralgia (PHN) or Peripheral Nerve Injury
MeSH Terms: conditions — Neuralgia, Postherpetic; Peripheral Nerve Injuries | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NT 201 (Experimental): Subcutaneous injections of up to 300 units NT 201 into the peripheral neuropathic pain area
  Interventions: Biological: IncobotulinumtoxinA
- Placebo (Placebo Comparator): Subcutaneous injections of placebo into the peripheral neuropathic pain area
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IncobotulinumtoxinA — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl)
  Other Names: Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins; NT 201
  Arms: NT 201
Biological: Placebo — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Arms: Placebo

SUMMARY:
In this clinical trial, participants with nerve pain after shingles or nerve injury will receive injections with NT 201 or placebo. The purpose is to measure the decrease of nerve pain with NT 201 compared to placebo.

Trial details include:

* Trial duration: 22-23 weeks;
* Treatment duration: 1 injection visit with a 20-week follow-up period;
* Visit frequency: 2 remote visits by phone/video call (1 week and 12 weeks after the injection); 2 on-site visits (6 weeks and 20 weeks after the injection).

ELIGIBILITY:
Inclusion Criteria:

* Chronic peripheral neuropathic pain that persists for at least 6 months by the time of the screening visit and is plausibly related to either an episode of herpes zoster or a peripheral nerve injury (caused by surgery or mechanical trauma).
* Documented diagnosis of either chronic neuropathic pain after peripheral nerve injury (i.e., postsurgical/post-traumatic neuropathic pain) or postherpetic neuralgia with at least probable level of certainty according to the NeuPSIG/IASP (Neuropathic Pain Special Interest Group / International Association on the Study of Pain) grading system.
* A score of at least 4 out of 10 points on the Neuropathic Pain 4 Questions (DN4) questionnaire.

Exclusion Criteria:

* Complex Regional Pain Syndrome Type 1 and Type 2.
* Any other painful condition or disease that requires treatment (only mild to moderate episodic migraine treated with triptans and/or non-steroidal anti- inflammatory drugs (NSAIDs), if any, is acceptable).
* Postsurgical/post-traumatic neuropathic pain due to amputation and/or phantom limb pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Weekly averages of changes from baseline in Average Daily Pain (ADP) intensity at Weeks 2 to 12. | Baseline to week 2 to 12

SECONDARY OUTCOMES:
Changes from baseline in Neuropathic Pain Symptom Inventory (NPSI) total score at Weeks 2 to 12 | Baseline to week 2 to 12
Incidence of treatment-emergent adverse events (TEAEs) related to study intervention as assessed by the investigator from intervention to end of study. | Baseline to week 20

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Therapeutics GmbH
Locations (31):
- Bulgaria (5):
  - Merz Investigational Site #3590004, Plovdiv
  - Merz Investigational Site #3590006, Sofia
  - Merz Investigational Site #3590005, Sofia
  - Merz Investigational Site #3590002, Sofia
  - Merz Investigational Site #3590003, Veliko Tarnovo
- France (3):
  - Merz Investigational Site #0330066, Boulogne-Billancourt
  - Merz Investigational Site #0330065, Limoges
  - Merz Investigational Site #0330067, Nîmes
- Germany (6):
  - Merz Investigational Site #0490174, Essen
  - Merz Investigational Site #0490386, Frankfurt
  - Merz Investigational Site #0490389, Hamburg
  - Merz Investigational Site #0490388, Kiel
  - Merz Investigational Site #0490219, Leipzig
  - Merz Investigational Site #0490387, Westerstede
- Hungary (3):
  - Merz Investigational Site #0360021, Budapest
  - Merz Investigational Site #0360020, Budapest
  - Merz Investigational Site #0360022, Budapest
- Poland (10):
  - Merz Investigational Site #0480113, Częstochowa
  - Merz Investigational Site #0480112, Gdynia
  - Merz Investigational Site #0480111, Katowice
  - Merz Investigational Site #0480115, Katowice
  - Merz Investigational Site #0480059, Krakow
  - Merz Investigational Site #0480114, Lublin
  - Merz Investigational Site #0480110, Poznan
  - Merz Investigational Site #0480109, Warsaw
  - Merz Investigational Site #0480107, Warsaw
  - Merz Investigational Site #0480108, Wroclaw
- Spain (4):
  - Merz Investigational Site #0340043, Barcelona
  - Merz Investigational Site #0340044, Córdoba
  - Merz Investigational Site #0340041, L'Hospitalet de Llobregat
  - Merz Investigational Site #0340042, Seville

IPD SHARING:
Plan to Share IPD: No